CLINICAL TRIAL: NCT01487564
Title: A Single-Dose, Open-Label Study to Evaluate the Pharmacokinetic Profile of OROS Hydromorphone in Healthy Adult Taiwanese Subjects Having Different Genotypes for the UGT2B7 Gene
Brief Title: Pharmacokinetic Profile of OROS Hydromorphone in Healthy Taiwanese Participants With Different Genotypes for the UGT2B7 Gene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR017701; 42801PAI1011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers; Pharmacokinetics; OROS Hydromorphone; Hydromorphone; Taiwan; UGT2B7 Gene
MeSH Terms: interventions — Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydromorphone 16 mg (Experimental)
  Interventions: Drug: Hydromorphone 16 mg

INTERVENTIONS:
Drug: Hydromorphone 16 mg — type= exact number, unit= mg, number= 16, format= tablet, route= oral use. One tablet of hydromorphone 16 mg.

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of OROS hydromorphone in healthy adult Taiwanese participants after the oral administration of a single 16 mg dose.

DETAILED DESCRIPTION:
This is a single-center, open-label (all people know the identity of the intervention), single-dose study in healthy adult Taiwanese participants. A minimum of 6 participants identified as having the UGT2B7 *2/*2 variant genotype and 12 participants identified as having the UGT2B7 *1/*1 wild type genotype will be included in the study. The study will explore the impact of genetic polymorphism in the UGT2B7 gene (occurrence of variants of this gene) on the pharmacokinetics (how the drug is absorbed in the body, distributed within the body, and how it is removed from the body over time) of OROS hydromorphone. This study consists of a screening phase followed by a 5-day open-label treatment phase. During the screening phase, a blood sample will be collected for a genetic test to confirm the presence of the UGT2B7 gene. During the study period, upon completion of a 12-hour overnight fast, participants will receive a single oral 16-mg dose of OROS hydromorphone in the morning of Day 1. Blood samples will be collected through 72 hours after dosing for the determination of plasma hydromorphone and hydromorphone 3-glucuronide concentrations. The safety and tolerability of 16-mg OROS hydromorphone will also be assessed. The total study duration for each participant is approximately 33 days.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the DNA analysis to confirm UGT2B7 genotype status
* Body mass index (BMI) between 18 and 25 kg/m², inclusive and a body weight of not less than 50 kg
* Participants must utilize a medically acceptable method of contraception throughout the entire study period and for 1 month after the study is completed
* Each participant will receive a naloxone challenge test for opioid dependency at screening. Only those participants who pass this challenge test will be allowed to continue in the study

Exclusion Criteria:

* History of or current clinically medical illness or any other condition that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Clinically significant abnormal values for hematology, clinical chemistry or urinalysis
* Clinically significant abnormal physical examination, vital signs or 12 lead electrocardiogram (ECG)
* Use of certain prescription or nonprescription medication, and consumption of products that may interfere with the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Plasma hydromorphone concentration | 20 time points up to 72 hours post-dose

SECONDARY OUTCOMES:
Plasma hydromorphone 3-glucuronide concentration | 20 time points up to 72 hours post-dose
Number of participants with adverse events as a measure of safety and tolerability | Approximately 33 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Development, L.L.C. Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Taipei, Taiwan